CLINICAL TRIAL: NCT00965094
Title: Efficacy and Safety of Certican® (Everolimus) in Combination With Myfortic® (EC-MPS, Enteric-coated Mycophenolate Sodium) After Early CNI Elimination Versus Myfortic® in Combination With Prograf® in Renal Transplant Recipients
Brief Title: Efficacy and Safety of Everolimus+EC-MPS After Early CNI Elimination vs EC-MPS +Tacrolimus in Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001AIL03
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Everolimus; Tacrolimus; Basiliximab; Mycophenolic Acid; Adrenal Cortex Hormones

ARMS (2):
- Everolimus (Experimental): At BL1, all study patients received induction therapy with basiliximab (Simulect®; 2x20mg on day 0 - 2 hours prior to transplantation, and on day 4 after transplantation) and commenced an immunosuppressive regimen consisting of MPA (Myfortic®; target dose: 1440 mg/day, which was also the maximum daily dose) + tacrolimus (Prograf®; based on C0-h levels; Table 9-2) and with corticosteroids. AT BL2 [Month 3 (+1 week) after transplantation], eligible patients were randomized, using living and cadaveric donation as stratum. Patients were switched to the CNI-free regimen. Everolimus was added to the patients immunosuppressive regimen and tacrolimus was removed successively.
  Interventions: Drug: Everolimus; Drug: Basiliximab; Drug: Enteric Coated Mycophenolate Sodium (EC-MPS); Drug: Corticosteroids
- Reference Therapy (Active Comparator): At BL1, all study patients received induction therapy with basiliximab (Simulect®; 2x20mg on day 0 - 2 hours prior to transplantation, and on day 4 after transplantation) and commenced an immunosuppressive regimen consisting of MPA (Myfortic®; target dose: 1440 mg/day, which was also the maximum daily dose) + tacrolimus (Prograf®; based on C0-h levels; Table 9-2) and with corticosteroids. AT BL2 [Month 3 (+1 week) after transplantation], eligible patients were randomized, using living and cadaveric donation as stratum. Patients continued on the prior immunosuppressive regimen consisting of MPA + tacrolimus with corticosteroids.
  Interventions: Drug: Tacrolimus (FK506); Drug: Basiliximab; Drug: Enteric Coated Mycophenolate Sodium (EC-MPS); Drug: Corticosteroids

INTERVENTIONS:
Drug: Everolimus — One tablet containing 0.25, 0.5mg or 0.75 mg. Initially 2 mg/day. Afterwards based on blood level (target 6-10 ng/mL)
  Other Names: Certican
  Arms: Everolimus
Drug: Tacrolimus (FK506) — Capsules 0.5 mg, 1 mg. Dosing according to blood level.
  Other Names: Prograf
  Arms: Reference Therapy
Drug: Basiliximab — One vial containing 20 mg lyophilisate. 2 x 20 mg [day 0 (2 hrs prior to Tx) and day 4 post Tx] to be applied as 10 sec. bolus injection, i.v.
  Other Names: Simulect
Drug: Enteric Coated Mycophenolate Sodium (EC-MPS) — One tablet containing 180 mg or 360 mg. 1440 mg/day (2x720 mg). If tolerated, dose reduction due to side effectis were possible (min. dose at BL@: 720 mg/day)
  Other Names: Myfortic
Drug: Corticosteroids — Used according to Israeli standards. A minimum dose of 5mg [prednisone, or equivalent, was used throughout the study period.

SUMMARY:
The primary objective of this trial is to show non-inferiority of a CNI-free regimen with respect to the renal function at Month 9 post Tx assessed by glomerular filtration rate - Nankivell method - as compared to the standard CNI-based regimen in de novo renal transplant patients.

ELIGIBILITY:
Inclusion criteria:

* Recipients of de novo cadaveric, living unrelated or living related kidney transplants
* Females capable of becoming pregnant must have a negative serum pregnancy test within 7 days prior to or at screening, and are required to practice an approved method of birth control for the duration of the study and for a period of 6 weeks following discontinuation of study medication, even where there has been a history of infertility.
* Patients who are willing and able to participate in the study and from whom written informed consent has been obtained.

Exclusion criteria:

* More than one previous renal transplantation
* Multi-organ recipients (e.g., kidney and pancreas) or previous transplant with any other organ, different from kidney
* Donor age: < 5 years or > 65 years
* Graft loss due to immunological reasons in the first year after transplantation (in case of secondary transplantation)
* Patients who had received an investigational drug within 4 weeks of the baseline period
* Patients who are recipients of A-B-O incompatible transplants or T cell cross-match positive transplants
* Patients with already existing antibodies against the HLA-type of the receiving transplant
* Patients with any known hypersensitivity to Simulect®, Certican®, mycophenolic acid, Prograf®, other drugs similar to Certican® (e.g., macrolides), or other components of the formulations.
* Patients who have received an investigational immunosuppressive drug within four weeks prior to study entry (Baseline visit 1)
* Patients with thrombocytopenia (platelets < 75,000/mm³), or an absolute neutrophil count of < 1,500/mm³ or leucopenia (leucocytes < 2,500/mm³), or hemoglobin < 6 g/dL
* Patients with preexisting lung disease (alveolitis, fibrosis) Patients with symptoms of significant somatic or mental illness. Inability to cooperate or communicate with the investigator, who are unlikely to comply with the study requirements, or who are unable to give informed consent
* Patients with a history of malignancy during the last five years, except squamous or basal cell carcinoma of the skin
* Patients who are HIV positive or Hepatitis B surface antigen positive or Hepatitis C virus positive. Recipients of organs from donors who test positive for Hepatitis B surface antigen or Hepatitis C are excluded.
* Evidence of severe liver disease (incl. abnormal liver enzyme profile, i.e. AST, ALT or total bilirubin > 3 times UNL)
* Females of childbearing potential who are planning to become pregnant, who are pregnant or lactating, and/or who are unwilling to use effective means of contraception (see also section 8.2)
* Presence of a clinically significant infection requiring continued therapy, severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus that in the opinion of the investigator would interfere with the appropriate conduct of the study
* Evidence of drug or alcohol abuse
* Patients receiving drugs known to interact with Tacrolimus and/or everolimus according to the list provided in Appendix 3 to this protocol.
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv

REFERENCES:
- [Background] Bemelman FJ, de Maar EF, Press RR, van Kan HJ, ten Berge IJ, Homan van der Heide JJ, de Fijter HW. Minimization of maintenance immunosuppression early after renal transplantation: an interim analysis. Transplantation. 2009 Aug 15;88(3):421-8. doi: 10.1097/TP.0b013e3181af1df6. PMID 19667948

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Everolimus | Reference Therapy
Started | 19 | 17
Completed | 14 | 16
Not Completed | 5 | 1
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled patient population included all patients who signed an informed consent regardless whether renal transplanation as performed or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus | Reference Therapy | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (13.4) | 49.6 (12.1) | 51.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Renal Function Assessed as Glomerula Filtration Rate (GFR) - Nankivell Method - 9 Months After Renal Transplantation (LOCF)
Description: The glomerular filtration rate (GFR) is the best clinical estimate of renal function in health and disease, and correlates well with the clinical severity of renal function disturbances. The GFR, calculated according to the Nankivell formula, was used as the primary outcome measure in this study. This equation has been validated in renal transplant patients against the true GFR measured by a radionuclide method and has been confirmed as a very accurate method to calculate the GFR in this specific population (Gaspari et al., 2004)GFR = 6.7 / Scr + BW / 4 - Surea / 2-100 / (height)² + C Scr = serum creatinine concentration expressed in mmol/L. BW = body weight in kg, Surea = serum urea in mmol/L and Height is expressed in meters.The Last Observation Carried Forward (LOCF) imputation technique was used for this analysis.
Time Frame: 9 months
Population: The ITT population comprised all randomized patients who received at least one dose of the study medications after randomization and had at least one post-baseline assessment of the primary efficacy variable (renal function based on Nankivell method).
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Groups:
- Reference Therapy: Control Arm: At BL1, all study patients received induction therapy with basiliximab (Simulect®; 2x20mg on day 0 - 2 hours prior to transplantation, and on day 4 after transplantation) and commenced an immunosuppressive regimen consisting of MPA (Myfortic®; target dose: 1440 mg/day, which was also the maximum daily dose) + tacrolimus (Prograf®; based on C0-h levels; Table 9-2) and with corticosteroids. AT BL2 [Month 3 (+1 week) after transplantation], eligible patients were randomized, using living and cadaveric donation as stratum. Patients continued on the prior immunosuppressive regimen consisting of MPA + tacrolimus with corticosteroids.
Arm/Group | Everolimus | Reference Therapy
Number analyzed (Participants) | 15 | 15
mL/min/1.73m^2 | 15.0 (10.3) | 16.6 (7.0)

2. Secondary Outcome: Assessment of GFR by the Cockcroft-Gault Method (LOCF)
Description: the GFR was also calculated using the Cockcroft-Gault method (Cockcroft and Gault 1976) and the Modification of Diet in Renal Disease (MDRD) method (Levey et al., 1999, Rodrigo et al., 2003; Pierrat et al., 2003).Cockcroft-Gault formula For men: GFR= (140-Age)X Body Weight[kg]/72X Serum Creatinine[mg/dl] For women: GFR= 0,85x(140-Age) x Body Weight[kg]/72x Serum Creatinine [mg/dl] The Last Observation Carried Forward (LOCF) imputation technique was used for this analysis.
Time Frame: 9 months
Population: The ITT population comprised all randomized patients who received at least one dose of the study medications after randomization and had at least one post-baseline assessment of the primary efficacy variable
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Everolimus | Reference Therapy
Number analyzed (Participants) | 15 | 15
mL/min | 72.6 (18.9) | 72.7 (20.5)

3. Secondary Outcome: Participants Who Had Occurrence of Biopsy Proven Acute Rejection, Graft Loss or Death.
Description: Biopsy-proven acute rejection was defined as a biopsy gradeed IA, IB, IIA, IIB, or III. The allograft was presumed to be lost if the patient started dialysis and was not able to subsequently be removed from dialysis. If the patient underwent a graft nephrectomy, then the day of nephrectomy was the day of graft loss.
Time Frame: 9 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Everolimus | Reference Therapy
Number analyzed (Participants) | 15 | 15
Participants
  No | 14 | 14
  Yes | 1 | 1

4. Secondary Outcome: Participants Who Had Occurrence of Treatment Failure.
Description: Treatment failure was defined as a composite endpoint of biopsy-proven acute rejection, graft loss, death, loss to follow up, discontinuation due to lack of efficacy or toxicity or conversion to another regimen.
Time Frame: 9 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Everolimus | Reference Therapy
Number analyzed (Participants) | 15 | 15
Participants
  No | 10 | 14
  Yes | 5 | 1

5. Secondary Outcome: Change in Renal Function (Creatinine Slope)
Description: X(slope)=(1/value of creatinine).
Time Frame: 3 months, 5 months, 7 months, 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl per month
Arm/Group | Everolimus | Reference Therapy
Number analyzed (Participants) | 15 | 15
mg/dl per month
  (ITT) Baseline 2: Month 3 N=15, 15 | 0.7 (0.1) | 0.7 (0.2)
  (ITT) Month 3 (1st week) N=15, 4 | 0.7 (0.2) | 0.8 (0.1)
  (ITT) Month 3 (2nd week) N=15, 4 | 0.8 (0.1) | 0.9 (0.2)
  (ITT) Month 3 (3rd week) N=13, 2 | 0.7 (0.1) | 0.9 (0.2)
  (ITT) Month 3 (4th week) N=12, 0* | 0.8 (0.1) | NA (NA) — No participants analyzed for this time point.
  (ITT) Month 5 N=14, 15 | 0.8 (0.2) | 0.7 (0.2)
  (ITT) Month 7 N=14, 14 | 0.7 (0.2) | 0.7 (0.2)
  (ITT) Month 9 N=11, 15 | 0.8 (0.2) | 0.8 (0.2)
  (PP) Baseline 2: Month 3 N=11, 15 | 0.7 (0.1) | 0.7 (0.2)
  (PP) Month 3 (first week) N=11, 4 | 0.7 (0.2) | 0.8 (0.1)
  (PP) Month 3 (second week) N=11, 4 | 0.8 (0.1) | 0.9 (0.2)
  (PP) Month 3 (third week) N=10, 2 | 0.7 (0.1) | 0.9 (0.2)
  (PP) Month 3 (fourth week) N=9, 0* | 0.8 (0.1) | NA (NA) — No participants analyzed for this time point.
  (PP) Month 5 N=11, 15 | 0.8 (0.2) | 0.7 (0.2)
  (PP) Month 7 N=11, 14 | 0.8 (0.2) | 0.7 (0.2)
  (PP) Month 9 N=11, 15 | 0.8 (0.2) | 0.8 (0.2)

ADVERSE EVENTS:
Arm/Group | Everolimus | Reference Therapy
Serious Adverse Events (participants affected / at risk) | 7/19 | 7/17
Other Adverse Events (participants affected / at risk) | 19/19 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=19) | Reference Therapy (N=17)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 2 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Craniotomy (Surgical and medical procedures) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=19) | Reference Therapy (N=17)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 5 | 1
Monocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Diabetes mellitus (Endocrine disorders) | 2 | 3
Hypercalcaemia (Endocrine disorders) | 1 | 0
Orbital oedema (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 2
Pyrexia (General disorders) | 3 | 0
Transplant rejection (Immune system disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Human polyomavirus infection (Infections and infestations) | 3 | 2
Infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 3
Blood lactate dehydrogenase (Investigations) | 4 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Epstein-Barr virus test positive (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 2 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Bladder pain (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 3
Glycosuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 6 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Bladder anastomosis (Surgical and medical procedures) | 0 | 1
Urethral repair (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.